CLINICAL TRIAL: NCT04714151
Title: A Phase III Confirmatory Study of K-877 Extended Release Tablet-A Multicenter, Active Controlled, Randomized, Double Blind, Parallel Group Controlled Trial in Patients With Dyslipidemia With High TG-
Brief Title: A Phase III Confirmatory Study of K-877 Extended Release Tablet
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kowa Company, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: K-877-ER-02
Record Dates: First submitted 2021-01-15; First posted 2021-01-19 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Dyslipidemias
MeSH Terms: conditions — Dyslipidemias | interventions — (R)-2-(3-((benzoxazol-2-yl-d4 (3-(4-methoxyphenoxy-d7)propyl)amino)methyl)phenoxy) butanoic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treatment A (Experimental): K-877 ER 0.2 mg/day (once daily)
  Interventions: Drug: K-877 ER 0.2 mg/day (once daily)
- Treatment B (Experimental): K-877 ER 0.4 mg/day (once daily)
  Interventions: Drug: K-877 ER 0.4 mg/day (once daily)
- Control A (Active Comparator): K-877 IR 0.2 mg/day (twice daily)
  Interventions: Drug: K-877 IR 0.2 mg/day (twice daily)

INTERVENTIONS:
Drug: K-877 ER 0.2 mg/day (once daily) — K-877 ER 0.2 mg tablet
  Other Names: Pemafibrate ER 0.2 mg/day (once daily)
  Arms: Treatment A
Drug: K-877 ER 0.4 mg/day (once daily) — K-877 ER 0.4 mg tablet
  Other Names: Pemafibrate ER 0.4 mg/day (once daily)
  Arms: Treatment B
Drug: K-877 IR 0.2 mg/day (twice daily) — K-877 IR 0.1 mg tablet
  Other Names: Pemafibrate IR 0.2 mg/day (twice daily)
  Arms: Control A

SUMMARY:
To investigate the efficacy and safety of K-877 Extended Release (ER) 0.2 mg/day or 0.4 mg/day (once daily) for 12 weeks in dyslipidemia, using K-877 Immediate Release (IR) 0.2 mg/day (twice daily) as a control.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with dyslipidemia had to be age 20 years or older at written informed consent
2. Patients who have received dietary or exercise guidance from 12 weeks or more prior to Screening
3. Patients with the fasting serum TG >= 200 mg/dL twice consecutively at Screening

Exclusion Criteria:

1. Patients with a fasting serum TG > 1000 mg/dL at Screening
2. Patients who require administration of prohibited drugs during the clinical trial period after written informed consent
3. Patients with uncontrolled thyroid disease
4. Patients with type 1 diabetes and uncontrolled diabetes [HbA1c(NGSP) >= 8.0 % at Screening]
5. Patients with uncontrolled hypertension (SBP >= 160 mmHg or DBP >= 100 mmHg)
6. Patients with an AST or ALT three times the upper limit at Screening
7. Patients with an CK five times the upper limit at Screening
8. Patients with cirrhosis or those with biliary obstruction
9. Patients with acute myocardial infarction within 3 months before obtaining informed consent
10. Patients with heart failure class III or higher according to NYHA cardiac function classification
11. Patients with malignant tumor or those who are judged to have a high risk of recurrence
12. Patients with a history of serious drug allergies (anaphylactic shock, etc.)
13. Pregnant women, lactating women, women planning to become pregnant or lactating during the study period, or pregnant women who do not use specific contraceptive methods
14. Patients who have collected 400 mL or more of whole blood within 16 weeks, or 200 mL or more of whole blood within 4 weeks, or blood samples (plasma and platelet components) within 2 weeks before Screening
15. Patients who have received K-877 (pemafibrate)
16. Patients who participate in other clinical trials at the time of written informed consent and who received medication or who have received clinical trials other than placebo for less than 16 weeks
17. Patients who have been determined inappropriate by the investigator, etc

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 356 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-09-25 (Actual); Study Completion 2021-09-25 (Actual)

PRIMARY OUTCOMES:
Efficacy : % change from baseline in fasting serum TG (mg/dL) | 4, 8, and 12 week after administration

SECONDARY OUTCOMES:
Efficacy : % change from baseline in fasting serum Total Cholesterol (mg/dL) | 4, 8, and 12 week after administration
Efficacy : % change from baseline in fasting serum LDL-C (mg/dL) | 4, 8, and 12 week after administration
Efficacy : % change from baseline in fasting serum HDL-C (mg/dL) | 4, 8, and 12 week after administration
Efficacy : % change from baseline in fasting serum non-HDL-C (mg/dL) | 4, 8, and 12 week after administration

CONTACTS AND LOCATIONS:
Locations (11):
- Japan (11):
  - Institute Medical Corporation Hitomikai Motomachi Takatsuka Naika Clinic, Kanagawa
  - Medical Corporation Heishinkai OCROM Clinic, Osaka
  - Dojinkinenkai Meiwa Hospital, Tokyo
  - Fukuwa Clinic, Tokyo
  - Ikebukuro Metropolitan Clinic, Tokyo
  - Medical Corp. Seikoukai New Medical Research System Clinic, Tokyo
  - Medical Corporation Asbo Tokyo Asbo Clinic, Tokyo
  - Medical Corporation Chiseikai Tokyo Center Clinic, Tokyo
  - Medical Corporation Heishinkai ToCROM Clinic, Tokyo
  - Medical Corporation Yuhokai Miho Clinic, Tokyo
  - Tokyo-Eki Center-building Clinic, Tokyo

REFERENCES:
- [Result] Arai H, Yamashita S, Araki E, Yokote K, Tanigawa R, Saito A, Yamasaki S, Suganami H, Ishibashi S. Efficacy and Safety of Pemafibrate Extended-Release Tablet: a Phase 3, Multicenter, Randomized, Double-Blind, Active-Controlled, Parallel-Group Comparison Trial. J Atheroscler Thromb. 2024 Nov 1;31(11):1517-1538. doi: 10.5551/jat.64677. Epub 2024 Apr 13. PMID 38616112